CLINICAL TRIAL: NCT05669092
Title: A Randomized, Controlled, Open-label, Multicenter, Phase III Trial of Anus-preservation in Low Rectal Adenocarcinoma Based on MMR/MSI Status(APRAM)
Brief Title: A Phase III Trial of Anus-preservation in Low Rectal Adenocarcinoma Based on MMR/MSI Status
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARTOnG 2201
Record Dates: First submitted 2022-11-28; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Toripalimab; Radiation
MeSH Terms: interventions — toripalimab; Capecitabine; Irinotecan; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A: dMMR/MSI-H patients (Experimental): patients will receive 12 cycles of PD-1 antibody
  Interventions: Drug: Toripalimab
- ARM B: dMMR/MSI-H patients (Experimental): patients will receive 5*5Gy short-course radiotherapy, followed by 12 cycles of PD-1 antibody
  Interventions: Drug: Toripalimab; Radiation: SCRT
- ARM C: pMMR/MSS patients (Experimental): patients will receive CRT followed by 6 cycles of XELIRI
  Interventions: Radiation: CRT; Drug: XELIRI
- ARM D: pMMR/MSS patients (Experimental): patients will receive CRT followed by 12 cycles of FOLFRINOX
  Interventions: Radiation: CRT; Drug: FOLFRINOX

INTERVENTIONS:
Drug: Toripalimab — 3mg/Kg iv d1q2w
  Other Names: PD-1inhibitor
  Arms: ARM A: dMMR/MSI-H patients; ARM B: dMMR/MSI-H patients
Radiation: CRT — IMRT 50Gy/25fx 625mg/m2 bid d1-5 qw Irinotecan:1、Full wild (GG+6/6): 80mg/m2/week for 5 times 2、Single site mutation (GG+6/7 or GA+6/6): 65mg/m2/week for 5 times 3、Double locus mutation (GG+7/7 or AA+6/6 or GA+6/7): 50mg/m2/week for the 1st, 2nd, 4th and 5th week for 4 times
  Other Names: LCRT
  Arms: ARM C: pMMR/MSS patients; ARM D: pMMR/MSS patients
Radiation: SCRT — 25Gy/5fx
  Other Names: short-course radiotherapy
  Arms: ARM B: dMMR/MSI-H patients
Drug: XELIRI — Capecitabine: 1000mg/m2 bid d1-14 Irinotecan: 200mg/m2 ivgtt d1 q3w
  Other Names: Capecitabine and Irinotecan
  Arms: ARM C: pMMR/MSS patients
Drug: FOLFRINOX — Irinotecan: 150mg/m2 ivgtt d1 (double locus mutation downregulated to 120mg/m2) Oxaliplatin: 85mg/m2 ivgtt d1 5-FU: 2400mg/m2 ivgtt 46h q2w
  Other Names: Irinotecan,Oxaliplatin and 5-FU
  Arms: ARM D: pMMR/MSS patients

SUMMARY:
pMMR/MSS and 32 dMMR/MSI-H patientspatients were planned to be enrolled. Patients with dMMR/MSI-H will be randomly assigned to the immunotherapy arm or short-course radiotherapy sequential immunotherapy arm; pMMR/MSS patients will receive capecitabine-irinotecan based concurrent radiotherapy before being randomly assigned to the XELIRI or FOLFRINOX arm.

The rate of complete response (sustained cCR for ≥ 1 year), long-term prognosis and adverse effects will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. pathological confirmed adenocarcinoma；
2. clinical stage T2-4 and/or N+，Not suitable for initial local excision to achieve radical treatment；
3. the distance from anal verge less than ≤ 5cm，or surgical evaluation concludes that direct surgical anal preservation is not possible without distance metastases；
4. age 18-70 years old, female and male；
5. Strong desire for anal preservation and ability to be closely monitored for at least 2 years after chemoradiotherapywith good compliance；
6. without distant metastases；
7. ECOG Performance status 0-1；
8. Detection of UGT1A1*6 and *28 gene status (for pMMR patients)；
9. Sufficient bone marrow reserve and physical capacity to receive consolidation chemotherapy after chemoradiotherapy (for pMMR patients)；
10. with good compliance；
11. signed the inform consen.

Exclusion Criteria:

1. pregnant or breastfeeding women；
2. Persons with a history of uncontrolled epilepsy, central nervous system disorders, or psychiatric disorders whose clinical severity, as judged by the investigator, may prevent the signing of informed consent or affect the patient's compliance with oral medications；
3. Difficult to achieve complete remission at the available level of evidence, such as: tumor largest diameter >10 cm; largest diameter of lateral lymph nodes >2 cm; baseline CEA >= 100; biopsy pathology with an indolent cell carcinoma component; tumor of circumferential narrowing type on anal finger examination, with inclusion decided by the judgment of the evaluation team if necessary；
4. Clinically significant (i.e., active) heart disease, such as symptomatic coronary artery disease, New York Heart Association (NYHA) class II or worse congestive heart failure or severe arrhythmias requiring pharmacological intervention, or a history of myocardial infarction within the last 12 months；
5. persons requiring immunosuppressive therapy for organ transplantation；
6. Persons with severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases；
7. Subjects with baseline routine blood and biochemical indicators do not meet the following criteria: hemoglobin ≥ 90g/L; absolute neutrophil count (ANC) ≥ 1.5×109/L; platelets ≥ 100×109/L; ALT, AST ≤ 2.5 times the upper limit of normal; ALP ≤ 2.5 times the upper limit of normal; serum total bilirubin < 1.5 times the upper limit of normal; serum creatinine < 1 times the upper limit of normal limit; serum albumin ≥30g/L；
8. Known to have dihydropyrimidine dehydrogenase (DPD) deficiency；
9. allergic to any investigational drug component.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate. | The status of cCR will be evaluated after the completion of neoadjuvant therapy.
  cCR ≥ 1 year.

SECONDARY OUTCOMES:
adverse effects rate. | From date of randomization until the date of death from any cause, assessed up to 5 years ] Rate of chemotherapy, radiotherapy and immunotherapy related adverse events.
  CTC 4.0 standard.
QoL | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using EORTC QLQ-C30 score
3 year local recurrence free survival rate | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months. ]
  Rate of 3 year local recurrence free survival
3 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months. ]
  Rate of 3 year disease free survival
3 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
Organ preservation | From date of randomization until the date of surgery
  TME-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengjiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Huang CY, Bai MH, Shen JW, Sun QQ, Feng YR, Chen QP, Mao W, Ju HX, Zhu J. Anus preservation in low rectal adenocarcinoma based on MMR/MSI status (APRAM): a study protocol for a randomised, controlled, open-label, multicentre phase III trial. BMC Cancer. 2024 Jan 10;24(1):57. doi: 10.1186/s12885-024-11829-2. PMID 38200410